CLINICAL TRIAL: NCT02980666
Title: A 24-week Safety, Efficacy, Pharmacodynamic, and Pharmacokinetic Study of Teduglutide in Japanese Pediatric Subjects, Aged 4 Months Through 15 Years, With Short Bowel Syndrome Who Are Dependent on Parenteral Support
Brief Title: Study in Japanese Pediatric Subjects With Short Bowel Syndrome (SBS) Who Are Dependent on Parenteral Support
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP633-302; 2020-005791-35 (EudraCT Number)
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Results first posted 2021-02-10 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2021-01

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Teduglutide (Experimental): Participants will receive teduglutide 0.05 milligram per kilogram per day (mg/kg/day) subcutaneous (SC) injection once daily for 24 weeks.
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — 0.05 mg/kg/day SC injection once daily for 24 weeks.

SUMMARY:
The purpose of this study is to determine if an investigational treatment (teduglutide) is safe and effective in Japanese children (age 4 months through 15 years of age) with SBS who are dependent on parenteral support. This study will also evaluate how teduglutide moves through the body (pharmacokinetics) and how it affects the body (pharmacodynamics).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by a parent or guardian prior to any study-related procedures
* When applicable, informed assent (as deemed appropriate by the Institutional Review Board) by the participant prior to any study-related procedures
* Male or female infant 4 to <12 months corrected gestational age or child or adolescent aged 1 year through 15 years
* Current history of SBS as a result of major intestinal resection (eg, due to necrotizing enterocolitis, midgut volvulus, intestinal atresia, or gastroschisis)
* Short bowel syndrome that requires PN/IV support that provides at least 30% of caloric and/or fluid/electrolyte needs
* Stable PN/IV support, defined as:

For infants 4 to <12 months corrected gestational age: Inability to significantly reduce PN/IV support, usually associated with minimal or no advance in enteral feeds (ie, 10% or less change in PN or advance in feeds) for at least 1 month prior to and during screening, as assessed by the investigator.

For children 1 to 15 years of age:

Inability to significantly reduce PN/IV support, usually associated with minimal or no advance in enteral feeds (ie, 10% or less change in PN or advance in feeds) for at least 3 months prior to and during screening, as assessed by the investigator.

Transient instability for events such as interruption of central access or treatment of sepsis is allowed if the PN/IV support returns to within 10% of baseline prior to the event.

- Sexually active female participants of childbearing potential must use medically acceptable methods of birth control during and for 4 weeks following the last dose of investigational product.

Exclusion Criteria:

* Participants who are not expected to be able to advance oral or tube feeding regimens
* Serial transverse enteroplasty or any other bowel lengthening procedure performed within 3 months of screening
* Known clinically significant untreated intestinal obstruction contributing to feeding intolerance and inability to reduce parenteral support
* Unstable absorption due to cystic fibrosis or other known DNA abnormalities (eg, Familial Adenomatous Polyposis, Fanconi-Bickel syndrome)
* Severe, known dysmotility syndrome such as pseudo-obstruction or persistent, severe, active gastroschisis-related dysmotility; that is the primary contributing factor to feeding intolerance and inability to reduce parenteral support, prior to screening. Dysmotility is defined as severe if it is expected to limit the advancement of enteral feeding.
* Evidence of clinically significant obstruction on the most recent upper GI series done within 6 months prior to screening.
* Major GI surgical intervention including significant intestinal resection within 3 months prior to screening (insertion of feeding tube, anastomotic ulcer repair, minor intestinal resections <=10 centimeter (cm), or endoscopic procedure is allowed)
* Unstable cardiac disease or congenital heart disease or cyanotic disease, with the exception of participants who had undergone ventricular or atrial septal defect repair, and patent ductus arteriosus (PDA) ligation
* History of cancer or clinically significant lymphoproliferative disease, not including resected cutaneous basal or squamous cell carcinoma, or in situ nonaggressive and surgically resected cancer. Participants with known cancer predisposition syndrome, such as juvenile polyposis or Beckwith-Wiedemann syndrome, or first degree relative with early onset of GI cancer (including hepatobiliary and pancreatic cancer) will also be excluded.
* Pregnant or lactating female participants
* Participation in a clinical study using an experimental drug (other than glutamine or Omegaven) within 3 months or 5.5 half-lives of the experimental drug, whichever is longer, prior to screening and for the duration of the study
* Previous use of teduglutide or native/synthetic GLP-2
* Previous use of glucagon-like peptide-1 analog or human growth hormone within 3 months prior to screening
* Previous use of octreotide or dipeptidyl peptidase-4 (DPP-4) inhibitors within 3 months prior to screening
* Participants with active Crohn's disease who had been treated with biological therapy (eg, antitumor necrosis factor [anti-TNF]) within the 6 months prior to the screening visit
* Participants with inflammatory bowel disease (IBD) who require chronic systemic immunosuppressant therapy that had been introduced or changed during the 3 months prior to screening
* More than 3 serious complications of SBS (eg, documented infection-related catheter sepsis, clots, bowel obstruction, severe water-electrolyte disturbances) within 3 months prior to the screening visit
* A serious complication that affects parenteral support requirements within 1 month prior to or during screening, excluding uncomplicated treatment of bacteremia, central line replacement/repair, or issues of similar magnitude in an otherwise stable participant
* Body weight < 5 kilogram (kg) at screening and baseline visits
* Signs of active, severe, or unstable clinically significant hepatic impairment during the screening period:

For infants 4 to <12 months corrected gestational age at least 2 of any of the following parameters:

1. International normalized ratio (INR) >1.5 not corrected with parenteral vitamin K
2. Platelet count <100×10^3/ (microliters)mcL due to portal hypertension
3. Presence of clinically significant gastric or esophageal varices
4. Documented cirrhosis
5. Persistent cholestasis defined as conjugated bilirubin >4 milligram per deciliter (mg/dL) (>68 micromoles per liter [mcmol/L]) over a 2 week period

For children 1 to 15 years of age:

1. Total bilirubin >= 2x upper limit of normal (ULN)
2. Aspartate aminotransferase (AST) >= 7x ULN
3. Alanine aminotransferase (ALT) >= 7x ULN

   * Signs of known continuous active or unstable, clinically significant renal dysfunction shown by results of an estimated glomerular filtration rate below 50 milliliter per minute (mL/min)/1.73 meter (m)^2
   * Parent(s)/guardian(s) and/or participants who are not capable of understanding or not willing to adhere to the study visit schedule and other protocol requirements
   * Unstable, clinically significant, active, untreated pancreatic or biliary disease
   * Any condition, disease, illness, or circumstance that in the investigator's opinion puts the participant at any undue risk, prevents completion of the study, or interferes with analysis of the study results.

Ages: 4 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (5):
- Japan (5):
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Kagoshima University, Kagoshima, Kagoshima-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Showa University, Shinagawa-ku, Tokyo-To

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites, …).

REFERENCES:
- [Derived] Chiba M, Masumoto K, Kaji T, Matsuura T, Morii M, Fagbemi A, Hill S, Pakarinen MP, Protheroe S, Urs A, Chen ST, Sakui S, Udagawa E, Wada M. Efficacy and Safety of Teduglutide in Infants and Children With Short Bowel Syndrome Dependent on Parenteral Support. J Pediatr Gastroenterol Nutr. 2023 Sep 1;77(3):339-346. doi: 10.1097/MPG.0000000000003867. Epub 2023 Jun 26. PMID 37364133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 centers in Japan between 13 January 2017 (first participant first visit) and 21 January 2020 (last participant last visit).
Pre-assignment Details: A total of 10 Japanese study participants were enrolled into the study, including 8 children ages 1 through 15 years of age and 2 infants aged 4 months through < 12 months of corrected gestational age. All the participants received treatment and completed the study.
Groups:
- Total Children (Aged: 1 to 15 Years): Participants aged from 1 through 15 years received teduglutide 0.05 milligram per kilogram per day (mg/kg/day) subcutaneous (SC) injection once daily for 24 weeks and completed the study at Week 28.
- Infants (Corrected Gestational Age: 4 to < 12 Months): Participants (Infants) from 4 through < 12 months of corrected gestational age received teduglutide 0.05 mg/kg/day SC injection once daily for 24 weeks and completed the study at Week 28.
Period: Overall Study
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Started | 8 | 2
Completed | 8 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population consisted of all participants who were enrolled into the study and met all eligible criteria for the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months) | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Customized [Count of Participants; unit: Participants] | 8 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Parenteral Support (PS) Volume at End of Treatment (EOT) Based on Dairy Data
Description: Absolute change from baseline in PS volume at EOT (up to Week 24) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period. Here, milliliter per kilogram per day is abbreviated as mL/kg/day.
Time Frame: Baseline, EOT (up to Week 24)
Population: ITT population consisted of all participants who were enrolled into the study and met all eligible criteria for the study.
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
mL/kg/day | -11.8 (8.47) | -26.2 (13.61)

2. Primary Outcome: Percent Change From Baseline in Parenteral Support (PS) Volume at End of Treatment (EOT) Based on Dairy Data
Description: Percent change from baseline in PS volume at EOT (up to Week 24) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: Baseline, EOT (up to Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Percent Change | -27.7 (31.79) | -26.7 (15.14)

3. Primary Outcome: Absolute Change From Baseline in Parenteral Support (PS) Caloric Intake at End of Treatment (EOT) Based on Dairy Data
Description: Absolute change from baseline in PS caloric intake at EOT (up to Week 24) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period. Here, kilo-calories per kilogram per day was abbreviated as (kcal/kg/day).
Time Frame: Baseline, EOT (up to Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
kcal/kg/day | -7.2 (8.70) | -13.8 (3.17)

4. Primary Outcome: Percent Change From Baseline in Parenteral Support (PS) Caloric Intake at End of Treatment (EOT) Based on Dairy Data
Description: Percent change from baseline in PS caloric intake at EOT (up to Week 24) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: Baseline, EOT (up to Week 24)
Population: ITT population consisted of all participants who were enrolled into the study and met all eligible criteria for this study.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Percent change | -26.2 (33.00) | -25.7 (2.73)

5. Primary Outcome: Absolute Change From Baseline in Plasma Citrulline at End of Treatment (EOT)
Description: Absolute change from baseline in plasma citrulline at EOT (up to Week 24) was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: Baseline, EOT (up to Week 24)
Population: ITT population consisted of all participants who were enrolled into the study and met all eligible criteria for this study. Data for this outcome measure was not planned to be collected and analyzed for infants.
Measure: Mean (Standard Deviation); unit: Micromoles per liter (mcmol/L)
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 0
Micromoles per liter (mcmol/L) | 3.2 (4.28) |

6. Primary Outcome: Percent Change From Baseline in Plasma Citrulline at End of Treatment (EOT)
Description: Percent change from baseline in plasma citrulline at EOT (up to Week 24) was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: Baseline, EOT (up to Week 24)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 0
Percent change | 39.2 (39.46) |

7. Primary Outcome: Absolute Change From Baseline in Enteral Nutritional (EN) Volume at End of Treatment (EOT) Based on Dairy Data
Description: Absolute change from baseline in EN volume at EOT (up to Week 24) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: Baseline, EOT (up to Week 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
mL/kg/day | 1.0 (7.14) | 0.6 (2.15)

8. Primary Outcome: Percent Change From Baseline in Enteral Nutritional (EN) Volume at End of Treatment (EOT) Based on Dairy Data
Description: Percent change from baseline in EN volume at EOT (up to Week 24) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: Baseline, EOT (up to Week 24)
Population: ITT population consisted of all participants who were enrolled into the study and met all eligible criteria for this study. Here, the number of participants analyzed refer to the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 4 | 2
Percent change | 53.1 (111.01) | -23.2 (36.89)

9. Primary Outcome: Absolute Change From Baseline in Enteral Nutritional (EN) Caloric Intake at End of Treatment (EOT) Based on Dairy Data
Description: Absolute change from baseline in EN caloric intake at EOT (up to Week 24) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: Baseline, EOT (up to Week 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
kcal/kg/day | 0.8 (5.60) | 0.3 (1.03)

10. Primary Outcome: Percent Change From Baseline in Enteral Nutritional (EN) Caloric Intake at End of Treatment (EOT) Based on Dairy Data
Description: Percent change from baseline in EN caloric intake at EOT (up to Week 24) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: Baseline, EOT (up to Week 24)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 4 | 2
Percent change | 56.8 (117.88) | -24.2 (38.06)

11. Primary Outcome: Number of Participants Who Achieved At Least 20 Percent (%) Reduction in Parenteral Support (PS) Volume at Week 24
Description: Number of participants who achieved at least 20% reduction in PS volume at Week 24 was reported.
Time Frame: Week 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 7 | 2
Participants | 4 | 1

12. Primary Outcome: Number of Participants Who Achieved At Least 20 Percent (%) Reduction in Parenteral Support (PS) Volume at End of Treatment (EOT)
Description: Number of participants who achieved at least 20% reduction in PS volume at EOT (up to Week 24) was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: EOT (up to Week 24)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Participants | 4 | 1

13. Primary Outcome: Number of Participants Who Achieved 100 Percent (%) Reduction in Complete Weaning of Parenteral Support (PS) Volume at End of Treatment (EOT)
Description: Number of participants who achieved at least 100% reduction in complete weaning of PS volume at EOT (up to Week 24) was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: EOT (up to Week 24)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Participants | 1 | 0

14. Primary Outcome: Number of Participants Who Achieved Greater Than or Equal to (>=) 20 Percent (%) Reduction in Parenteral Support (PS) Volume at Week 28
Description: Number of participants who achieved >= 20% reduction in PS volume at Week 28 was reported.
Time Frame: Week 28
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Participants | 3 | 1

15. Primary Outcome: Absolute Change From End of Treatment (EOT) in Parenteral Support (PS) Volume at End of Study (EOS) Based on Dairy Data
Description: Absolute change from EOT (up to Week 24) in PS volume at EOS (up to Week 28) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: EOT (up to Week 24), EOS (up to Week 28)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
mL/kg/day | 3.9 (7.06) | -3.8 (0.67)

16. Primary Outcome: Percent Change From End of Treatment (EOT) in Parenteral Support (PS) Volume at End of Study (EOS) Based on Dairy Data
Description: Percent change from EOT (up to Week 24) in PS volume at EOS (up to Week 28) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: EOT (up to Week 24), EOS (up to Week 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 7 | 2
Percent change | 9.8 (19.59) | -5.5 (2.35)

17. Primary Outcome: Absolute Change From End of Treatment (EOT) in Parenteral Support (PS) Caloric Intake at End of Study (EOS) Based on Dairy Data
Description: Absolute change from EOT (up to Week 24) in PS caloric intake at EOS (up to Week 28) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: EOT (up to Week 24), EOS (up to Week 28)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
kcal/kg/day | 0.5 (6.16) | -4.0 (1.38)

18. Primary Outcome: Percent Change From End of Treatment (EOT) in Parenteral Support (PS) Caloric Intake at End of Study (EOS) Based on Dairy Data
Description: Percent change from EOT (up to Week 24) in PS caloric intake at EOS (up to Week 28) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: EOT (up to Week 24), EOS (up to Week 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 7 | 2
Percent change | 3.5 (19.17) | -10.3 (4.40)

19. Primary Outcome: Absolute Change From End of Treatment (EOT) in Plasma Citrulline at End of Study (EOS)
Description: Absolute change from EOT (up to Week 24) in plasma citrulline at EOS (up to Week 28) was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: EOT (up to Week 24), EOS (up to Week 28)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Micromoles (mcM)
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 0
Micromoles (mcM) | -2.9 (2.87) |

20. Primary Outcome: Percent Change From End of Treatment (EOT) in Plasma Citrulline at End of Study (EOS)
Description: Percent change from EOT (up to Week 24) in plasma citrulline at EOS (up to Week 28) was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: EOT (up to Week 24), EOS (up to Week 28)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 0
Percent change | -20.0 (24.16) |

21. Primary Outcome: Absolute Change From End of Treatment (EOT) in Enteral Nutritional (EN) Volume at End of Study (EOS) Based on Dairy Data
Description: Absolute change from EOT (up to Week 24) in EN volume at EOS (up to Week 28) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: EOT (up to Week 24), EOS (up to Week 28)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
mL/kg/day | -1.5 (3.24) | -2.8 (3.98)

22. Primary Outcome: Percent Change From End of Treatment (EOT) in Enteral Nutritional (EN) Volume at End of Study (EOS) Based on Dairy Data
Description: Percent change from EOT (up to Week 24) in EN volume at EOS (up to Week 28) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: EOT (up to Week 24), EOS (up to Week 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 4 | 2
Percent change | -22.1 (28.06) | -1.4 (8.25)

23. Primary Outcome: Absolute Change From End of Treatment (EOT) in Enteral Nutritional (EN) Caloric Intake at End of Study (EOS) Based on Dairy Data
Description: Absolute change from EOT (up to Week 24) in EN caloric intake at EOS (up to Week 28) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: EOT (up to Week 24), EOS (up to Week 28)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
kcal/kg/day | -1.1 (2.64) | -1.4 (1.97)

24. Primary Outcome: Percent Change From End of Treatment (EOT) in Enteral Nutritional (EN) Caloric Intake at End of Study (EOS) Based on Dairy Data
Description: Percent change from EOT (up to Week 24) in EN caloric intake at EOS (up to Week 28) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: EOT (up to Week 24), EOS (up to Week 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 4 | 2
Percent change | -22.1 (28.16) | -3.0 (6.03)

25. Primary Outcome: Absolute Change From Baseline in Number of Hours Per Day of Parenteral Support (PS) Usage at End of Treatment (EOT) Based on Dairy Data
Description: Absolute change from baseline in number of hours per day of PS Usage at EOT (up to Week 24) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: Baseline, EOT (up to Week 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hours per day (hours/day)
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Hours per day (hours/day) | -2.1 (4.16) | 0.0 (0.00)

26. Primary Outcome: Absolute Change From Baseline in Number of Days Per Week of Parenteral Support (PS) Usage at End of Treatment (EOT) Based on Dairy Data
Description: Absolute change from baseline in number of days per Week of PS usage at EOT (up to Week 24) based on dairy data was reported. EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period.
Time Frame: Baseline, EOT (up to Week 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days per week
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Days per week | -0.9 (2.47) | 0.0 (0.00)

27. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs were defined as any AEs whose onset occurred, severity worsened, or intensity increased after receiving the investigational product.
Time Frame: From start of study drug administration up to EOS (up to Week 28)
Population: Safety population consisted of all participants in the ITT population who received at least 1 administration of investigational product with any safety follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Participants | 8 | 2

28. Primary Outcome: Change From Baseline in Body Weight for Age Z-score at Week 28
Description: Body weight was measured using age Z-score. A Z-score was defined as the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in body weight for age Z-score at Week 28 was reported.
Time Frame: Baseline, Week 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Z-score | 0.177 (0.3625) | 2.332 (1.1503)

29. Primary Outcome: Change From Baseline in Height for Age Z-score at Week 28
Description: Height was measured using age Z-score. A Z-score was defined as the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-score at Week 28 was reported.
Time Frame: Baseline, Week 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Z-score | 0.024 (0.4841) | 1.056 (0.6968)

30. Primary Outcome: Change From Baseline in Head Circumference for Age Z-score at Week 28
Description: Head circumference was measured using age Z-score. A Z-score was defined as the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in head circumference for age Z-score at Week 28 was reported.
Time Frame: Baseline, Week 28
Population: Safety population consisted of all participants in the ITT population who received at least 1 administration of investigational product with any safety follow-up. Data for this outcome measure was not planned to be collected and analyzed for Total Children (Aged: 1 to 15 Years).
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 2
Z-score |  | 1.559 (0.6116)

31. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Reported as Treatment Emergent Adverse Events (TEAEs)
Description: Vital sign assessments included pulse rate, blood pressure, or body temperature. Number of participants with clinically significant changes in vital signs by the investigator were recorded as TEAEs.
Time Frame: From start of study drug administration up to EOS (up to Week 28)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Participants | 0 | 0

32. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Reported as Treatment Emergent Adverse Events (TEAEs)
Description: 12-lead ECG was performed. Any change in ECG assessments which were deemed to be clinically significant changes were recorded as TEAEs.
Time Frame: From start of study drug administration up to EOS (up to Week 28)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Participants | 0 | 0

33. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Reported as Treatment Emergent Adverse Events (TEAEs)
Description: Clinical laboratory assessments included biochemistry, hematology, coagulation, urinalysis. The number of participants with clinically significant laboratory abnormalities were reported as TEAEs.
Time Frame: From start of study drug administration up to EOS (up to Week 28)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Participants | 0 | 0

34. Primary Outcome: Change From Baseline in the Average Urine Output at Week 28
Description: Average urine output was recorded in measured volume at Week 28 was recorded.
Time Frame: Baseline, Week 28
Population: Safety population consisted of all participants in the ITT population who received at least 1 administration of investigational product with any safety follow-up. Here, the number of participants analyzed refer to the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 7 | 1
mL/kg/day | -22.317 (34.8252) | -48.879 (NA) — Standard deviation was not estimated as only single participant was analyzed.

35. Primary Outcome: Change From Baseline in the Fecal Output at Week 28
Description: Change from baseline in the fecal output (Average number of stools per day) at Week 28 was recorded.
Time Frame: Baseline, Week 28
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Average number of stools per day
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 7 | 1
Average number of stools per day | -0.64 (1.547) | 2.50 (NA) — Standard deviation was not estimated as only single participant was analyzed.

36. Primary Outcome: Number of Participants With Positive Specific Antibodies to Teduglutide
Description: Number of participants with positive specific antibodies to teduglutide were used to summarize the presence of antibodies.
Time Frame: From start of study drug administration up to EOS (up to Week 28)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 2
Participants | 1 | 2

37. Primary Outcome: Number of Participants With Clinically Significant Abnormal Findings in Gastrointestinal (GI) Specific Testing
Description: GI specific testing included colonoscopy or sigmoidoscopy, abdominal ultrasound, fecal occult blood testing, upper GI series with small bowel follow-through (UGI/SBFT). EOT was defined as the last available measurement after the date of first dose during the 24-week treatment period. Number of participants with clinically significant abnormal findings in gastrointestinal specific testing were reported.
Time Frame: Baseline, EOT (up to Week 24)
Population: Safety population consisted of all participants in the ITT population who received at least 1 administration of investigational product with any safety follow-up. Data for this outcome was not planned to be collected and analyzed for infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 8 | 0
Participants | 0 |

38. Primary Outcome: Area Under the Concentration-time Curve at Steady State (AUCtau,ss) of Teduglutide in Plasma
Description: Since only 2 sparse pharmacokinetics (PK) samples were collected during the study, PK parameters were not estimated and analyzed using this study samples. Therefore, no PK parameters were reported in this study.
Time Frame: Baseline: Pre-dose, 1, 6 hours post-dose; Week 4: Pre-dose, 2, 4 hours post-dose
Population: Since only 2 sparse PK samples were collected during the study, PK parameters were not estimated and analyzed using this study samples. Therefore, no PK parameters were reported in this study.
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 0

39. Primary Outcome: Maximum Plasma Concentration at Steady-state (Cmax,ss) of Teduglutide in Plasma
Description: Since only 2 sparse PK samples were collected during the study, PK parameters were not estimated and analyzed using this study samples. Therefore, no PK parameters were reported in this study.
Time Frame: Baseline: Pre-dose, 1, 6 hours post-dose; Week 4: Pre-dose, 2, 4 hours post-dose
Population: as for outcome 38
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 0

40. Primary Outcome: Minimum Plasma Concentration at Steady-state (Cmin.ss) of Teduglutide in Plasma
Description: as for outcome 39
Time Frame: Baseline: Pre-dose, 1, 6 hours post-dose; Week 4: Pre-dose, 2, 4 hours post-dose
Population: as for outcome 38
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 0

41. Primary Outcome: Time to Reach Maximum Observed Drug Concentration (Tmax) of Teduglutide in Plasma
Description: as for outcome 39
Time Frame: Baseline: Pre-dose, 1, 6 hours post-dose; Week 4: Pre-dose, 2, 4 hours post-dose
Population: as for outcome 38
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 0

42. Primary Outcome: Terminal-Phase Half-life (t1/2) of Teduglutide in Plasma
Description: as for outcome 39
Time Frame: Baseline: Pre-dose, 1, 6 hours post-dose; Week 4: Pre-dose, 2, 4 hours post-dose
Population: as for outcome 38
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 0

43. Primary Outcome: Apparent Clearance (CL/F) of Teduglutide
Description: as for outcome 39
Time Frame: Baseline: Pre-dose, 1, 6 hours post-dose; Week 4: Pre-dose, 2, 4 hours post-dose
Population: as for outcome 38
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 0

44. Primary Outcome: Apparent Volume of Distribution (V[Lambda z]/F) of Teduglutide
Description: as for outcome 39
Time Frame: Baseline: Pre-dose, 1, 6 hours post-dose; Week 4: Pre-dose, 2, 4 hours post-dose
Population: as for outcome 38
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to end of the study (up to Week 28)
Groups:
- Total Children (Aged: 1 - 15 Years): Participants aged from 1 through 15 years received teduglutide 0.05 mg/kg/day SC injection once daily for 24 weeks and completed the study at Week 28.
Arm/Group | Total Children (Aged: 1 - 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/2
Serious Adverse Events (participants affected / at risk) | 6/8 | 2/2
Other Adverse Events (participants affected / at risk) | 8/8 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Children (Aged: 1 - 15 Years) (N=8) | Infants (Corrected Gestational Age: 4 to < 12 Months) (N=2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (4)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 3 (4) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2)
Device damage (Product Issues) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Children (Aged: 1 - 15 Years) (N=8) | Infants (Corrected Gestational Age: 4 to < 12 Months) (N=2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site granuloma (General disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 2 (9) | 0 (0)
Injection site erythema (General disorders) | 3 (12) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 1 (4) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 6 (6) | 1 (1)
Frostbite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperzincaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Device damage (Product Issues) | 2 (2) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT02980666/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT02980666/SAP_001.pdf